CLINICAL TRIAL: NCT01593514
Title: A Single Centre, Open-label, Randomised Clinical Study to Investigate Meningococcal Serogroup A and C Saccharide Specific B Cell Responses in Adult Volunteers to One of Three Regimens of Meningococcal ACWY Conjugate Vaccine or Meningococcal ACWY Polysaccharide Vaccine Priming Doses Followed by a Booster Dose of the Meningococcal ACWY Conjugate Vaccine
Brief Title: Understanding the Immune Response to Two Different Meningitis Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OVG 2012/02
Record Dates: First submitted 2012-04-19; First posted 2012-05-08 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Meningitis; Meningococcal Disease; Septicaemia
Keywords: Vaccines; Meningitis; Meningococcal
MeSH Terms: conditions — Meningitis; Meningococcal Infections; Toxemia | interventions — Meningococcal Vaccines; lactitol; halofantrine; Polysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 Conjugate-conjugate (Active Comparator): Group I will receive 2 doses of the MenACWY-CRM conjugate vaccine (Novartis Vaccines) given 1 month apart. All vaccine doses are 0.5ml and will be administered intramuscularly into the deltoid.
  Interventions: Biological: MenACWY-CRM conjugate vaccine (Menveo, Novartis)
- Group 2 Polysaccharide-conjugate (Experimental): Group II will receive one full dose of MenACWY-PS polysaccharide vaccine meningococcal vaccine, followed by one dose of MenACWY-CRM conjugate vaccine given 1 month later.
  0.5 mL of MenACWY-PS vaccine will be administered subcutaneously and 0.5 mL of the MenACWY-CRM vaccine will be administered intramuscularly into the deltoid.
  Interventions: Biological: MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis)
- Group 3 Polysaccharide (subcutaneously)-conjugate (Experimental): Group III will receive a full dose of MenACWY-PS polysaccharide vaccine meningococcal vaccine subcutaneously, followed by one dose of MenACWY-CRM conjugate vaccine given 1 month later.
  Interventions: Biological: MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis); Biological: 1/5th dose MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis)
- Group 4: 1/5th dose Polysaccharide:conjugate (Experimental): Group IV will receive one fifth dose of MenACWY-PS polysaccharide vaccine meningococcal vaccine, followed by one dose of MenACWY-CRM conjugate vaccine given 1 month later.
  0.1 mL of MenACWY-PS vaccine will be administered IM and 0.5 mL of the MenACWY-CRM vaccine will be administered intramuscularly into the deltoid.
  Interventions: Biological: Polysaccharide (subcutaneously)-conjugate

INTERVENTIONS:
Biological: MenACWY-CRM conjugate vaccine (Menveo, Novartis) — The MenACWY-CRM conjugate vaccine (Menveo, Novartis) is obtained by extemporaneous mixing just before injection of the lyophilized MenA component to be reconstituted with the MenCWY component. This vaccine is to be administered intramuscularly.
  Arms: Group 1 Conjugate-conjugate
Biological: MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis) — The MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) is obtained by reconstituting the purified ACWY polysaccharides with the 0.5 ml water for injection. This vaccine should be administered subcutaneously.The MenACWY-CRM conjugate vaccine (Menveo, Novartis) is obtained by extemporaneous mixing just before injection of the lyophilized MenA component to be reconstituted with the MenCWY component. This vaccine is to be administered intramuscularly.
  Arms: Group 2 Polysaccharide-conjugate
Biological: MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis) — The MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) is obtained by reconstituting the purified ACWY polysaccharides with the 0.5 ml water for injection. This vaccine should be administered subcutaneously.The MenACWY-CRM conjugate vaccine (Menveo, Novartis) is obtained by extemporaneous mixing just before injection of the lyophilized MenA component to be reconstituted with the MenCWY component. This vaccine is to be administered intramuscularly.
  Arms: Group 3 Polysaccharide (subcutaneously)-conjugate
Biological: 1/5th dose MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) and MenACWY-CRM conjugate vaccine (Menveo, Novartis) — To obtain the one-fifth dose of MenACWY-PS, 0.5ml of a full dose of MenACWY-PS will be reconstituted, and then 0.4ml will be discarded prior to subcutaneous injection. The MenACWY-CRM conjugate vaccine (Menveo, Novartis) is obtained by extemporaneous mixing just before injection of the lyophilized MenA component to be reconstituted with the MenCWY component. This vaccine is to be administered intramuscularly.
  Arms: Group 3 Polysaccharide (subcutaneously)-conjugate
Biological: Polysaccharide (subcutaneously)-conjugate — The MenACWY-PS polysaccharide vaccine, ( ACWYVax, GSK) is obtained by reconstituting the purified ACWY polysaccharides with the 0.5 ml water for injection.The MenACWY-CRM conjugate vaccine (Menveo, Novartis) is obtained by extemporaneous mixing just before injection of the lyophilized MenA component to be reconstituted with the MenCWY component. This vaccine is to be administered subcutaneously
  Arms: Group 4: 1/5th dose Polysaccharide:conjugate

SUMMARY:
The bacterium (germ) Neisseria meningitidis causes meningitis and blood poisoning. N meningitidis is classified into different serogroups (types), based on its outer polysaccharide (carbohydrate) capsule. Serogroups A,B,C,W & Y are responsible for the vast majority of meningococcal disease worldwide.

Older vaccines against types A,C,W & Y contain part of the polysaccharide capsule of the germ. However, these polysaccharide vaccines do not provide long-term protection against disease and are less effective in young children, the group most at risk of meningococcal disease. Newer "conjugate" ACWY vaccines attach a polysaccharide to a protein carrier - these provoke a good response in young children and can provide long-term protection.

White blood cells called B cells produce antibodies, which are the main components of protection against meningococcal disease. Although many studies have investigated the immune response to these vaccines in different age groups by measuring specific antibodies, there is limited information about the B cells underlying such an immune response. Several different subsets (populations) of B cells exist in the blood. Previous studies by the investigators group suggest that different numbers of B cells are produced in response to each vaccine type. However, little is understood about which subset of B cell is important for antibody production in response to these polysaccharide or conjugate vaccines.

This study aims to provide detailed information on the immune response to meningococcal vaccines by investigating the appearance of B cells and their subsets in the blood after vaccination with the polysaccharide and conjugate vaccines. These observations will help us understand how polysaccharide and conjugate vaccines stimulate the immune system in different ways. This knowledge will help in the development of new vaccines that are effective across all age groups.

The investigators aim to recruit 20 adults aged 30-70 from Oxfordshire. The study will be funded by the Oxford Vaccine Group.

DETAILED DESCRIPTION:
EPIDEMIOLOGY

Neisseria meningitidis is a globally important cause of meningitis and septicaemia. The polysaccharide capsule is an important virulence factor in causing invasive disease. The serogroup of a meningococcal strain is determined by the biochemical composition of the polysaccharide capsule. There are 13 diverse polysaccharide capsules but only A, B, C, W and Y commonly cause invasive infections. In particular serogroups A,C,W, & Y account for >70% of meningococcal disease in North America, serogroups B & C are responsible for the vast majority of disease in Europe and Serogroup A causes cyclical meningitis epidemics in the African meningitis belt, including the recent outbreak in 2009/2010.

Given the rapid progression and serious sequelae of meningococcal disease, primary prevention is vital and this is most effectively achieved by vaccination. In the absence of a serogroup B vaccine, quadrivalent vaccines against serogroups ACW & Y represent the broadest mechanism of control of meningococcal disease worldwide. Protection induced by these vaccines relies on anti-capsular polysaccharide antibodies.

MENINGOCOCCAL POLYSACCHARIDE AND CONJUGATE VACCINES

Polysaccharide ACWY vaccines consist of pure capsular polysaccharide from each of the four serogroups and have been in widespread use since the late 1970's. However, in common with polysaccharide vaccines against other encapsulated bacteria, meningococcal polysaccharide vaccines are poorly immunogenic in young children, do not provoke long lasting immune responses[5] and may not reduce nasopharyngeal carriage. Newer conjugate vaccines consist of capsular oligosaccharides chemically linked to a protein carrier. Conjugation of a polysaccharide to a protein carrier allows the recruitment of cognate T cell help with subsequent exposure to antigen provoking a potentiated antibody response and immunological memory.

This study aims to investigate novel aspects of the B cell immune responses to meningococcal polysaccharide and conjugate vaccines. To achieve this, we will administer a quadrivalent ACWY polysaccharide vaccine (MenACWY-PS), and a quadrivalent ACWY conjugate vaccine (MenACWY-CRM) containing capsular oligosaccharides of serogroups A, C, W-135 & Y conjugated to a CRM197 mutant diphtheria toxoid carrier to adult volunteers. Each of these vaccines contains different amounts of capsular antigen (see Table 1). The polysaccharide vaccine has 50µg of polysaccharide from each of the 4 serogroups, while the conjugate has 10µg of A and 5µg of each of C, W & Y.

A recent trial using MenACWY-PS and MenACWY-CRM conducted by the Oxford Vaccine Group (Understanding the Immune Response to Meningitis Vaccines, OXREC 09/H0606/20, Eudract 2007-001349-17) showed preliminary evidence of a difference in B cell responses to polysaccharide and conjugate meningococcal vaccines. However, a confounding factor in interpreting the data from this trial has been the difference in the amount of capsular antigen contained in each of the two types of vaccine used in the study.

Full dose MenACWY-PS Polysaccharide vaccine has 50µg each of MenA, MenC,MenW and MenY capsular antigen. MenACWY-CRM Conjugate vaccine contains 10µg of MenA capsular antigen and 5µg each of MenC, MenW and MenY.

The current study is designed to compare both the full dose MenACWY-PS and a 1/5th dose of MenACWY-PS (which contains 10µg of each serogroup) to a full dose of MenACWY-CRM. This will differentiate between a polysaccharide dose-dependent response and a true polysaccharide vaccine vs. conjugate vaccine response. In particular, we aim to investigate the thymus dependent or thymus independent nature of the immune response to polysaccharide and conjugate meningococcal vaccines respectively.

THYMUS INDEPENDENT AND THYMUS DEPENDENT IMMUNE RESPONSES

Thymus independent (TI) antigens are defined by their ability to induce immune responses in T-cell deficient or athymic mice. In common with other high molecular weight molecules with repetitive structures, polysaccharide vaccine antigens are further classified as Type 2 TI antigens. The repetitive polysaccharide epitopes cross-link the BCR of antigen specific B cells, triggering activation signals and stimulating proliferation and differentiation into antibody-secreting plasma cells. The absence of T cell help precludes the generation of memory B cells.

TI responses are thought to be largely mediated by marginal zone B cells (MZB), which mature in the marginal zone of the spleen. This compartment is poorly developed in children under two years of age, which results in an ineffective anti-polysaccharide immune response in this age group. Murine studies have revealed an important role for a further subset of mature B cells, B1b cells, in adaptive immunity . Unlike the development of conventional B cell memory, which requires the formation of germinal centres and T cells, the development of B1b cell-mediated long-lasting antibody responses occur independently of T cell- help.

In contrast, conjugate vaccines act as thymus dependent (TD) antigens. Binding of the polysaccharide moiety to antigen specific B cell receptors allows uptake of the polysaccharide protein conjugate and processing via the classical MHC class II pathway. Peptides derived from the carrier protein are presented to cognate CD4+ T helper cells, which provide signals for further B cell differentiation.

TD responses are mediated by follicular B cells (FOB), with generation of antibody secreting plasma cells and memory B cells, capable of responding to further specific antigenic challenge[10]. Recent work conducted at the Oxford Vaccine Group suggests that pneumococcal polysaccharide and conjugate vaccines induce B1b and FOB cells, respectively. This study will investigate whether this also holds true for meningococcal conjugate and polysaccharide vaccines. This will be done by analysing the different populations of B cells produced in response to the full dose polysaccharide vaccine, 1/5th polysaccharide vaccine and conjugate vaccine using novel immunological techniques developed in our laboratories.

HYPORESPONSIVENESS

Vaccine-induced hyporesponsiveness is the inability to mount a booster response of at least the same magnitude as that produced to the priming dose. Previous vaccination with meningococcal polysaccharide vaccine has been shown to impair antibody responses to subsequent meningococcal polysaccharide or conjugate vaccines. The design of this study will allow investigation of the phenomenon of polysaccharide induced hyporesponsiveness in quadrivalent meningococcal vaccines at the level of memory B cell and plasma cell responses.

SEROGROUP A

Unlike the sialic acid based polysaccharide capsules of serogroups B, C, W-135 & Y, serogroup A meningococcal capsules are composed of N-acetyl mannosamine phosphate. Plain serogroup A polysaccharide vaccines show unexpected immunogenicity in young infants.These results suggest that perhaps due to its chemical structure, group A polysaccharide may not be handled by the immune system as a classic TI antigen. This study will test the hypothesis that follicular B cells are produced in response to the serogroup A component of MenACWY-PS, and by contrast, marginal zone or B1b cells are produced in response to the serogroup C component of the same vaccine. This study will also test the hypothesis that follicular B cells are produced in response to serogroups A and C components of MenACWY-CRM.

ANTIBODY REPERTOIRE

The human humoral response is anticipatory; potential specific antibody exists prior to encountering the extensive collection of antigen encountered over the lifetime of an individual. The basis for this diverse repertoire is the multiple gene segments comprising the variable region of the antibody molecule. The potential for each V D & J segment to combine randomly introduces combinatorial diversity to the repertoire. During rearrangement, further nucleotides may be added to or removed from the junction of the gene segments, termed junctional diversity. Furthermore, during maturation of the antibody response, somatic hypermutation of the variable region occurs during B cell proliferation in the germinal centres. This underlies the increase in antibody affinity in secondary responses to antigen. These mechanisms help create a potential repertoire of up to 1016 antibody molecules.

Previous studies have shown that the human humoral response to specific antigens is restricted in diversity within the individual and across populations with a limited number of antibody encoding variable region genes being utilised. These studies have relied on traditional vector cloning and Sanger sequencing of rearranged heavy chain loci of single cells, and are limited in the scope of their analysis of potential repertoire.

Massive parallel sequencing and emulsion PCR are powerful new tools enabling large scale DNA sequencing with the potential to simultaneously sequence up to one million reads per run. These techniques have been applied to look at the potential antibody repertoire in zebrafish, the human antibody repertoire in specific B cell subsets[20] and to assess clonality of leukaemoid cells. This study aims to compare the VDJ repertoire in memory B cell populations before and after polysaccharide and conjugate ACWY vaccination.

ANALYSIS OF GENETIC INFLUENCES ON THE IMMUNE RESPONSE

A further aspect to be assessed in this study is the impact of genetic factors on the response to immunisation. Twin studies on several vaccines including measles, mumps and rubella, have shown high heritability of vaccine antibody responses. Some genetic associations have already been identified between genes of the adaptive and innate immune response and some vaccines, for example human leukocyte antigen (HLA) alleles and measles antibody responses and IL-1β polymorphisms and hepatitis B vaccine responses. These studies have been small scale and based on single candidate genes and the extent to which genetic variation contributes to vaccine responses remains poorly understood. Insight into which genetic variants affect responses to specific vaccines will help identify the critical immune pathways leading to protection after vaccination and lead to the production of more effective vaccines. In addition, the identification of genes that may play important roles in wild-type infection will allow a better understanding of disease pathogenesis, which in turn may lead to the development of novel therapies

The blood samples obtained in this study provide a source of DNA can then contribute to a DNA bank pooling samples from multiple different Oxford Vaccine Group studies. These DNA samples can then be used for genome wide analysis of the genetic factors influencing the host response to the vaccines received in the relevant studies. This DNA extraction and storage will only occur with the specific consent of participants, and DNA will not be analysed for any other purpose than to assess factors influencing the immune response to vaccines. Serum left over from separation of the cellular plug for DNA extraction will also be stored and further immunological assays such as the quantification of functional antibody by serum bactericidal activity may also be performed on them.

SUMMARY

This study aims to investigate in detail aspects of the B cell response to conjugate and polysaccharide quadrivalent meningococcal vaccines in healthy adults using a variety of novel laboratory methods.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following conditions in order to be enrolled:

* Between 30 and 70 years of age inclusive;
* Willing and able to give informed consent for participation after the nature of the study has been explained;
* In good health as determined by:

medical history history-directed physical examination clinical judgment of the investigator

* Able (in the Investigators opinion) and willing to comply with all study requirements including be available for all the visits scheduled in the study;
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

Participants with any of the following conditions or characteristics will be excluded from study enrolment:

* Prior receipt of a meningococcal vaccine;
* Prior laboratory confirmed disease caused by N meningitides;
* Prior history of any anaphylactic shock, asthma, urticarial or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
* Known or suspected autoimmune disease or impairment /alteration of immune function resulting from (for example):

  * Receipt of immunostimulants
  * Congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding year or long-term systemic corticosteroid therapy (prednisolone or equivalent for more than two consecutive weeks within the past 3 months).
* Suspected or known HIV infection or HIV related disease;
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months
* Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* Any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
* Participation in another clinical trial investigating a vaccine, a drug, a medical device, or a medical procedure;
* Pregnancy as confirmed by a positive pregnancy test ;
* Concurrent breast-feeding.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
phenotype of meningococcal serogroup A specific B cells | 7 days after immunisation
  The phenotype of meningococcal serogroup A specific B cells will be observed at day 7 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose quadrivalent meningococcal polysaccharide vaccine and quadrivalent meningococcal conjugate vaccine by Fluorescent Activated Cell Sorting (FACS) analysis. This will be performed at the laboratories of the Oxford Vaccine Group, University of Oxford.

SECONDARY OUTCOMES:
The phenotype of meningococcal serogroup C specific B cells | 28 days after immunisation
  The phenotype of meningococcal serogroup C specific B cells will be observed at day 28 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose quadrivalent meningococcal polysaccharide vaccine and quadrivalent meningococcal conjugate vaccine using flow cytometry.
The measurement of meningococcal serogroup A and C specific memory B cells | 28 days after immunisation
  The measurement of meningococcal serogroup A and C specific memory B cells at day 28 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose Quadrivalent meningococcal polysaccharide vaccine or quadrivalent meningococcal conjugate vaccine, and after the booster immunisation with the conjugate vaccine.
The phenotype of meningococcal serogroup A specific B cells | 28 days after immunisation
  The phenotype of meningococcal serogroup A specific B cells will be observed at day 28 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose quadrivalent meningococcal polysaccharide vaccine and quadrivalent meningococcal conjugate vaccine by Fluorescent Activated Cell Sorting (FACS) analysis. This will be performed at the laboratories of the Oxford Vaccine Group, University of Oxford.
The phenotype of meningococcal serogroup C specific B cells | 7 days after immunisation
  The phenotype of meningococcal serogroup C specific B cells will be observed at day 7 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose quadrivalent meningococcal polysaccharide vaccine and quadrivalent meningococcal conjugate vaccine using flow cytometry.
The measurement of meningococcal serogroup A and C specific plasma cells | 7 days after immunisation
  The measurement of meningococcal serogroup A and C specific plasma cells at day 7 following the initial immunisation with full dose quadrivalent meningococcal polysaccharide vaccine, 1/5th dose Quadrivalent meningococcal polysaccharide vaccine or quadrivalent meningococcal conjugate vaccine, and after the booster immunisation with the conjugate vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, BA, MBBS, FRCPCH, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Vaccine Group, Oxford, Oxfordshire, United Kingdom